CLINICAL TRIAL: NCT06568432
Title: Effect of C-reactive Protein and Serum Amyloid a Point-of-care Testing on Antibiotic Prescribing for Acute Respiratory-tract Infections At Village Clinics in China: a Study Protocol for a Cluster Randomised Controlled Trial
Brief Title: Effect of CRP and SAA Point-of-care Testing on Antibiotic Prescribing for Acute Respiratory-tract Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Xiaoxv Yin, PhD, Professor and Head of Social Medicne and Health Management Department, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HuazhongU20240822
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Antibiotic Prescribing for Acute Respiratory-tract Infections
Keywords: point-of-care testing; acute respiratory-tract infections; primary care facilities; Antibiotic prescription

STUDY DESIGN:
Intervention Model Description: In parallel arm design, subjects are randomized to one or more study arms and each study arm will be allocated a different intervention. After randomization each subject stays in their assigned treatment arm for the duration of the study.
  Subjects receive the same treatment throughout the trial. The results are then compared.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The control group will not have any intervention, as the control (usual care)
- Intervention group (Experimental): CRP&SAA POCT will be provided in 20 village clinics in the intervention group and additional physician training on the use of CRP&SAA POCT will be provided (including centralized and unified training, distribution of physician training manuals and desk reminders)
  Interventions: Device: CRP+SAA POCT

INTERVENTIONS:
Device: CRP+SAA POCT — CRP+SAA POCT will be provided in 20 village clinics in the intervention group
  Arms: Intervention group

SUMMARY:
The study was a practical, cluster-randomized controlled trial to evaluate the impact of CRP and SAA point-of-care testing (CRP&SAA POCT) on antibiotic prescribing in patients with acute respiratory-tract infections (ARI) at primary care facilities in rural China.

DETAILED DESCRIPTION:
The study was a practical, cluster-randomized controlled trial to evaluate the impact of CRP and SAA point-of-care testing (CRP&SAA POCT) on antibiotic prescribing in patients with acute respiratory-tract infections (ARI) at primary care facilities in rural China. The study includes two arms, in which CRP&SAA POCT will be provided in 20 village clinics in the intervention arm. Additional physician training on the use of CRP&SAA POCT (including centralized training, distribution of physician training manuals, and desk reminders) and patient education sheets (to help patients understand the help of CRP&SAA POCT in guiding their care) will also be provided；The control arm will not receive any intervention and will serve as the control (usual care). The primary outcome is the proportion of patients who are diagnosed with ARIs and prescribed antibiotics during their initial visit (defined as no prescription record at the current institution within the preceding 14 days) in both study arms.

ELIGIBILITY:
Eligibility criteria for clusters Village clinics with an annual outpatient volume exceeding 2000, an average of 10 or more patients per week presenting with ARIs, and licensed prescribers are considered eligible for selection for the intervention. Annual outpatient prescriptions and average weekly visits for ARIs will be verified by obtaining prescription data from all village clinics for the previous year, as documented in the information section of the local health board.

Eligibility criteria for participants The target population of this study included (1) patients of all ages diagnosed by a village doctor with ARIs (including upper and lower respiratory infections); and (2) patients who present with ≥1 acute respiratory symptoms (including cough, rhinitis (sneezing, nasal congestion or runny nose), sore throat, shortness of breath, wheezing or abnormal auscultation). Patients with non-respiratory diseases or those with severe clinical symptoms requiring referral to a higher-level institution are excluded from the target population.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19424 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the proportion of patients who are diagnosed with ARIs and prescribed antibiotics during their initial visit (defined as no prescription record at the current institution within the preceding 14 days) in both study arms. | between the start of intervention and 6 months of follow-up
  This outcome serves as the primary indicator, reflecting the overall impact of a comprehensive intervention based on CRP&SAA POCT in guiding antibiotic use for patients with ARIs. Since most self-limiting ARIs are caused by viral infections that do not require antibiotic treatment, the decline in antibiotic prescribing rates suggests that village doctors are prescribing antibiotics more judiciously. The selection of this outcome is both feasible and reliable within the context of village clinics in China. This is due to the transition of prescriptions from traditional paper documents to electronic storage, which allows for the proper preservation of prescription records, thereby ensuring data integrity and traceability.

SECONDARY OUTCOMES:
The proportion of multiple antibiotic prescriptions in the intervention and control arms. | between the start of intervention and 6 months of follow-up
  The proportion of multiple antibiotic prescriptions in the intervention and control arms (specifically, the proportion of ARI prescriptions that include two or more antibiotics).
The intravenously injected antibiotic prescription rate | between the start of intervention and 6 months of follow-up
  The intravenously injected antibiotic prescription rate (the proportion that contain any antibiotics delivered by intravenous injection)
The proportion containing any Traditional Chinese Medicines. | between the start of intervention and 6 months of follow-up
  The investigators included the proportion of participants using any form of Traditional Chinese Medicines as a secondary outcome. In the investigators' previous trials, the investigators observed an increase in the use of Traditional Chinese Medicines, possibly as an alternative to antibiotics.
The mean cost of an ARI prescription | between the start of intervention and 6 months of follow-up
  The mean cost of an ARI prescription, based on the cost of any medicines.
The mean cost of a consultation | between the start of intervention and 6 months of follow-up
  The mean cost of a consultation, based on all costs including medicines, tests and the consultation.

CONTACTS AND LOCATIONS:
Locations (1):
- 40 Village Clinics, Xiantao, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu M, Zhang Z, Ge E, Xie CX, Bai X, Zhu Y, Kuang G, Li J, Wang J, Wei X, Yin X. Effect of C-reactive protein and serum amyloid A point-of-care testing on antibiotic prescribing for acute respiratory-tract infections at village clinics in China: A study protocol for a cluster randomised controlled trial. PLoS One. 2025 Sep 8;20(9):e0331646. doi: 10.1371/journal.pone.0331646. eCollection 2025. PMID 40920832